CLINICAL TRIAL: NCT00351754
Title: Detection of Pulmonary Embolism Comparing Isovue-370 and Visipaque 320 Using 64-Slice Multi-Detector Computed Tomographic Angiography
Brief Title: Detection of Pulmonary Embolism With CECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IOP 106
Record Dates: First submitted 2006-06-30; First posted 2006-07-13 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Iopamidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Isovue

SUMMARY:
To compare the vascular enhancement of the two contrast agents in pulmonary Multi-detector CTA

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 yrs or older
* With suspected PE
* Referred for MDCTA of pulmonary arteries
* Signed informed consent

Exclusion Criteria:

* Pregnant and lactating females
* History of hypersensitivity to iodinated contrast agents
* Hyperthyroidism or pheochromocytoma
* Severe CHF
* Renal impairment
* Weight greater than 300 lbs
* Pacemaker
* Swan Ganz catheter
* Defibrillator or other intrathoracic metallic vascular device
* Received an investigational compound within 30 days of being in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-07; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Hounsfield Units (HU) measured at various levels of pulmonary arteries

SECONDARY OUTCOMES:
Presence of artifacts; global enhancement

CONTACTS AND LOCATIONS:
Overall Officials: Steve Sireci, M.D., Study Director — Bracco Diagnostics
Locations (1):
- Bracco Diagnostics, Inc., Princeton, New Jersey, United States